CLINICAL TRIAL: NCT06881459
Title: The Effect of Oxytocin on the Alpha Cell Response to Hypoglycaemia in Patients With Type 1 Diabetes
Acronym: GLOXY-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, Associate Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GLOXY-2; H-24080204 (Other: The Danish Health Research Ethics Committee system)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, single-arm study. Each participant goes through two experimental days in a randomized order, acting as their own controls
Who Masked: Participant, Investigator
Masking Description: The randomized order of infusions is blinded to both participant and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infusion of placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Infusion of oxytocin (Experimental): Infusion of oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Other: Placebo — Saline
  Arms: Infusion of placebo
Drug: Oxytocin — Oxytocin
  Arms: Infusion of oxytocin

SUMMARY:
Investigating the effect of oxytocin on pancreatic endocrine functions by determining glucagon secretion during hypoglycemia in participants with type 1 diabetes.

DETAILED DESCRIPTION:
Glucagonotropic effects of oxytocin will be examined in 16 participants with type 1 diabetes, during a hypoglycaemic clamp with concomitant intravenous infusion of synthetic oxytocin or placebo in a randomised, double-blinded design. This will determine the effect of oxytocin on the glucagon response to hypoglycemia. Additional changes in plasma/serum concentrations of insulin, C-peptide, glucose, glucose-dependent insulinotropic polypeptid (GIP) and glucagon-like peptide 1 (GLP-1) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index from 19 to 30 kg/m2
* T1D (diagnosed according to the criteria of the World Health Organization) with HbA1c <69 mmol/mol (<8.5%)
* T1D duration of 3-30 years
* C-peptide negative (stimulated C-peptide ≤ 100 pmol/l)
* Treatment with a stable basal-bolus or insulin pump regimen for ≥3 months

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Liver disease (alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times normal values) or present hepatobiliary and/or gastrointestinal disorder(s)
* Kidney disease (serum creatinine above normal range)
* Late microvascular complications except mild non-proliferative retinopathy
* Regular tobacco smoking or use of other nicotine-containing products
* Long QTc on electrocardiogram (ECG) at screening (≥0.45 seconds)
* Pituitary gland disease
* Treatment with any glucose-lowering drugs besides insulin
* Any ongoing medication or physical or psychological condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Glucagon secretion | From time 30 to time 90 minutes
  Glucagon secretion, measured as the difference in plasma glucagon response to hypoglycaemia (as assessed by baseline subtracted area under curve (bsAUC)) during the hypoglycaemic clamp, between study days with oxytocin and with placebo

SECONDARY OUTCOMES:
Glucagon during recovery | From time 90 minutes to time 135 minutes
  measured as difference in glucagon bsAUC in the recovery phase
Glucagon during the entire period | From time 0 minutes to time 135 minutes
  measured as difference in glucagon bsAUC in the intire period
Glucose infusion | From time 0 minutes to time 135 minutes
  measured as the total amount of glucose infused
Insulin | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of insulin between study days
c-peptide | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of c-peptide between study days
Epinephrine | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of epinephrine between study days
Norepinephrine | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of norepinephrine between study days
Cortisol | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of cortisol between study days
Cross-linked C-telopeptide of type I collagen( CTX) | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of CTX between study days
Procollagen type I N-terminal propeptide (P1NP) | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of P1NP between study days
Growth Hormone (GH) | From time 0 minutes to time 135 minutes
  measured as the difference in circulating levels of GH between study days

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No